CLINICAL TRIAL: NCT04205110
Title: Development and Validation of a Fast, Semi-Automated Hybrid Imaging Platform to Assess Coronary Atherosclerotic Plaque Morphology, Endothelial Shear Stress and Arterial Inflammation: A Proof of Principle Study (VALID-PET-CT)
Acronym: VALID-PET-CT
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19/LO/1086
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stable Angina; Coronary Artery Disease
Keywords: Intravascular Ultrasound; Near Infrared Spectroscopy; Positron Emission Tomography
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET-CT — PET-CT compared to intravascular imaging for assessment of atherosclerotic plaques in stable angina patients

SUMMARY:
Imaging the inside of coronary arteries (intravascular imaging) offers great insight into the assessment and treatment of coronary artery disease. Over time, substances such as fat, cholesterol and calcium can build up into 'plaques' in the arteries, causing narrowings or even blockages. These plaques can also rupture, causing cardiovascular events such as heart attacks or strokes. By using ultrasound and infrared technology, intravascular imaging can help assess these plaques, however this is an invasive technique involving angiography. Plaque composition, structure and stability can be affected by inflammation and the stress that the arteries are under. The investigators have pioneered novel minimally-invasive methods for modelling arterial stress using computed tomography coronary angiography (CTCA), as well as imaging coronary arterial inflammation using a positron emission tomography (PET) scan. Before embarking upon a large-scale clinical outcome study to determine whether these novel methods can improve risk prediction, the aim is to perform a proof-of-principle study to further develop our methodology for hybrid image analysis, and to validate this technique against high-resolution intravascular imaging as a surrogate marker of histology.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥40
2. Stable angina, defined as typical symptoms with evidence of reversible ischemia in non-invasive test and/or documented obstructive coronary artery disease on coronary angiography
3. Patient that is willing and can provide written informed consent.

Exclusion Criteria

1. Acute coronary syndrome within <3 months
2. Pregnancy
3. Estimated glomerular filtration rate (eGFR) <60ml/min/1.73m²
4. Previous bypass surgery
5. Decompensated heart failure, or left ventricular ejection fraction less than 30%
6. Patient allergic to contrast or cannot receive treatment with aspirin, heparin, or thienopyridines
7. Anticipated life expectancy <2 years
8. Flow limiting coronary artery disease in the proximal segments of all the 3 epicardial coronaries
9. History of heart transplantation
10. Patient that requires surgical revascularization
11. Extensive coronary artery disease (i.e., multiple chronic total occlusions) or tortuous coronary anatomy that does not allow assessment of the

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable angina patients with known coronary artery disease referred for further invasive assessment as part of routine clincal care
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Faesibility of co-registration of CTCA and PET-CT data | 12 months
  All studied vessels will be dividen into 3 mm segments and the CTCA and PET-CT studies will be co-registered electronically. The faesibility of this will be reported

SECONDARY OUTCOMES:
Comparing PET-CT, CTCA and intravascular imaging: plaque volume | 12 months
  The co-registered vessels will be dividen into 3 mm segments and the CTCA and PET-CT data will be compared with intravascular imaging as gold standard to compare estimations of plaque burden expressed as volume
Comparing PET-CT, CTCA and intravascular imaging: plaque composition | 12 months
  The co-registered vessels will be dividen into 3 mm segments and the CTCA and PET-CT data will be compared with intravascular imaging as gold standard to compare estimations of plaque composition (reported as type of plaque)
Comparing PET-CT, CTCA and intravascular imaging: haemodynamic forces | 12 months
  The co-registered vessels will be divided into 3 mm segments and the CTCA and PET-CT data will be compared with intravascular imaging as gold standard to compare estimations of haemodynamic forces including plaque and endothelial shear stress
Comparing PET-CT, CTCA and intravascular imaging: presence of inflammation | 12 months
  The co-registered vessels will be divided into 3 mm segments and the CTCA and PET-CT data will be compared with intravascular imaging as gold standard to compare assessment of markers of inflammation and vulnerability in the plaques identified

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No